CLINICAL TRIAL: NCT05419206
Title: Department of Infectious Disease and Clinical Microbiology
Brief Title: The Relationship Between CMV* Reactivation and Anti-cytokine Treatment in Critical COVID-19 Patients
Acronym: Cytomegalovir
Status: Completed | Type: Observational
Sponsor: Ramazan Gozukucuk (Other)
Responsible Party: Sponsor-Investigator, Ramazan Gozukucuk, Assos Prof Dr, Hisar Intercontinental Hospital
Organization: Hisar Intercontinental Hospital (Other)
Other Study IDs: HisarIH-101
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: COVID-19, Cytomegalovirus (CMV), Tocilizumab, Anakinra, Mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 cases with anticytokine therapy: Considering the use of anti-cytokines in these patients, it was found that 53 received tocilizumab, 27 received anakinra, and 10 received both. CMV DNA was positive in 38 (22.7%) of the patients included in the study. CMV positivity was found to be significantly higher in 90 patients (31.11%) compared to 77 patients (16.88%) who did not receive anti-cytokine treatment (p:0.033)
  Interventions: Diagnostic Test: CMV DNA analysis
- COVID-19 cases without anticytokine therapy: MV positivity was found to be significantly higher in 90 patients (31.11%) compared to 77 patients (16.88%) who did not receive anti-cytokine treatment (p:0.033)
  Interventions: Diagnostic Test: CMV DNA analysis

INTERVENTIONS:
Diagnostic Test: CMV DNA analysis — CMV DNA quantitative viral load levels were studied

SUMMARY:
The risk of secondary infection is high in critical patients hospitalized with the diagnosis of COVID-19. Immunosuppressive treatments are commonly used in critical COVID-19 patients, and immune dysfunction and CMV reactivation can be unnoticed in these patients.

DETAILED DESCRIPTION:
The records of critical patients were reviewed retrospectively. Whether these patients used tocilizumab and/or anakinra and their relationship with CMV reactivation were examined. Furthermore, the relationship between CMV reactivation and mortality and anti-cytokine treatment in patients was also examined. A total of 167 critical COVID-19 patients were included in the study, of which 38 (22.7%) were found to be CMV DNA positive. CMV positivity in patients treated with anti-cytokines (31.11%) was found to be significantly higher than in patients who were not treated with it (16.88%) (p:0.033). There was no significant difference in viral load levels (p:0.513). Furthermore, it was determined that anti-cytokine treatment significantly decreased mortality (p: 0.003) and that there was no significant relationship between CMV reactivation and mortality (p: 0.399). Even though CMV reactivation was high in critical COVID-19 patients who received anti-cytokine treatment, positive developments in morbidity and mortality were observed with early diagnosis and effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients over the age of 18 diagnosed with COVID-19 and patients followed in the intensive care unit.

Exclusion Criteria:

* Patients under the age of 18 with a mild/moderate course of COVID-19,
* CMV PCR positive before anti-cytokine treatment,
* patients who underwent hematopoietic stem cell transplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The mean age of the patients was 59.2 (26-91 years), 63.7 years for women, and 58.6 years for men. The study included 167 critical and/or intensive care patients, 24 of whom were female (14%), and 143 of whom were men.
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
The relationship between CMV reactivation and anti-cytokine treatment | 2020-2021
  CMV positivity was found to be significantly higher in who receive anti-cytokine treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hisar Hospital Intercontinental, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
published data

REFERENCES:
- [Derived] Gozukucuk R, Kilic HH. The relationship between CMV reactivation, anti-cytokine treatment and mortality in critical COVID-19 patients. Pak J Med Sci. 2023 Sep-Oct;39(5):1286-1290. doi: 10.12669/pjms.39.5.7301. PMID 37680795